CLINICAL TRIAL: NCT00495768
Title: Reducing Depressive Symptoms During HCV Therapy: A Randomized Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Texas Veterans Health Care System (U.S. Federal Agency)
Responsible Party: Dr, Stephen L. Stern, Audie L. Murphy VA Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 034-0013-391
Record Dates: First submitted 2007-07-02; First posted 2007-07-03 (Estimated); Last update posted 2007-12-14 (Estimated); Status verified 2007-12

CONDITIONS: Hepatitis C; Depression
Keywords: Hepatitis C; HCV; Depression; Interferons; Ribavirin
MeSH Terms: conditions — Hepatitis C; Depression | interventions — Sensitivity Training Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Behavioral: Group Training — Participants will be trained in techniques that are useful to cope with possible side effects of treatment, such as: keeping a journal (expressive writing), breathing exercises, cognitive behavioral therapy, mindfulness meditation, and exercise.

SUMMARY:
The purpose of this study is to conduct a randomized controlled trial of an 8-visit non-pharmacologic group intervention in reducing the severity of depressive symptoms in veterans who receive IFN and ribavirin for the treatment of Hepatitis C. We hypothesize that over the first 6 months of treatment with IFN and ribavirin for the 45 patients who receive the 8-visit intervention early in the course of treatment in addition to usual care (experimental group) will have lower scores on the CES-D, a standard depression rating scale, than the 45 patients who receive only usual care (control group).

DETAILED DESCRIPTION:
In this study, subjects will be randomly assigned (by chance, like the flipping of a coin) to one of two study groups. Half the subjects will be assigned to a training program, which will consist of 8 sessions over a period of 8 weeks in which they will be instructed in cognitive therapy ( a method of identifying and "talk back" to one's negative thoughts) and a variety of other stress-reducing techniques. The other half will be assigned to a control groups, which will no receive instruction in cognitive therapy or the other stress-reducing techniques. All subjects, both those in the training program and in the control group, will receive the usual care for hepatitis C that all patients in the Hepatology Clinic receive. All subjects will also be asked to participate in 6 testing visits over the course of the study. The first testing visit will last about 3 hours, which the others will last between 1 1/2 and 2 hours. Subjects will alo be interviewed by telephone about their personal and family medical and psychiatric history. This will take about an hour.

ELIGIBILITY:
Inclusion Criteria:

* Eligibility and interest in treatment for chronic HCV (Hepatitis C).
* Absence of co-infection of HIV or Hepatitis B.
* Age 25-68 years old.
* No treatment with IFN (interferon-alpha) in the past 6 months.
* Residence within a 3-hour drive of the clinic.

Exclusion Criteria:

* Patients must be willing to undergo treatment with PEG-interferon and ribavirin. They must be aware of the side effects of treatment and be motivated to self-administer the medications and come to regularly scheduled appointments.
* Patients with diabetes mellitus must have good glycemic control. Their Hgb A1 c must be <8.0%.
* Patients must not have an active malignancy.
* If patients have a history of severe psychiatric illness or are found to have one by screening with the CES-D, a psychiatrist must approve treatment. If the psychiatric problem is minor, it can be managed by the primary care physician or hepatitis C provider.
* Autoimmune disease, such as autoimmune hepatitis, systemic lupus erythematosis, or sarcoidosis, is a contraindication to treatment.
* Active alcohol or intravenous drug use is a contraindication to treatment.
* Patients with a seizure disorder muct be seizure-free for 6 months prior to treatment.
* Patients with a known history of coronary heart disease are excluded.
* Patients with complications of cirrhosis may not be treatment candidates. Those who have a platelet count of <50,000, large esophageal varices (grade 3-4), uncontrolled ascites, or uncontrolled encephalopathy are excluded.
* Patients with severe mental retardation or dementia are excluded because of difficulty in self-administration of medication and in tolerating the side effects.
* The patient and partner much agree to observe strict contraception to avoid pregnancy, since the medication is fetotoxic up to 6 months after treatment completion.

Ages: 25 Years to 68 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2004-07; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Patients in the experimental group will have less of an increase in their HAM-D score over the first 6 months of treatment; score on a depression rating scale at study visits 1-5. | Two years

SECONDARY OUTCOMES:
Patients in the experimental group will have less of an increase in their PHQ-9 score over the first 6 months of treatment; score on a rating scale at study visits 1-5. | Two years
Patients in the experimental group will have less of an increase in their BDI score over the first 6 months of treatment; score on a rating scale at study visits 1-5. | Two years
Fewer patients in the experimental group will have developed a major depressive episode over the first 6 months of treatment; score on MDD module (MINI)at study visits 1-5. | Two years
Patients in the experimental group will have less of a decline in their self-rated general health (item #1 of the SF-36) over the first 6 months of treatment. | Two years
Patients in the experimental group will have less of an increase in self-rated irritability (item #6 of the BSI ) over the first 6 months of treatment. | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Stephen L. Stern, M.D., Principal Investigator — South Texas Veterans Hospital, Audie Murphy Division & the University of Texas Health Science Center at San Antonio
Locations (1):
- South Texas Veterans Healthcare System, Audie Murphy Division, San Antonio, Texas, United States

REFERENCES:
- [Background] Akaike H. A new look at the statistical identification model. IEEE, Tranactions Auto Control 1974;19:716-23
- [Background] Alter MJ, Kruszon-Moran D, Nainan OV, McQuillan GM, Gao F, Moyer LA, Kaslow RA, Margolis HS. The prevalence of hepatitis C virus infection in the United States, 1988 through 1994. N Engl J Med. 1999 Aug 19;341(8):556-62. doi: 10.1056/NEJM199908193410802. PMID 10451460
- [Background] American Psychiatric Association. Diagnostic and Statistical Manual of Mental Disorders, 4th Edition, Text Revision (DSM-IV-TR), Washington, DC, 2000.
- [Background] Capuron L, Gumnick JF, Musselman DL, Lawson DH, Reemsnyder A, Nemeroff CB, Miller AH. Neurobehavioral effects of interferon-alpha in cancer patients: phenomenology and paroxetine responsiveness of symptom dimensions. Neuropsychopharmacology. 2002 May;26(5):643-52. doi: 10.1016/S0893-133X(01)00407-9. PMID 11927189
- [Background] Hauser P, Khosla J, Aurora H, Laurin J, Kling MA, Hill J, Gulati M, Thornton AJ, Schultz RL, Valentine AD, Meyers CA, Howell CD. A prospective study of the incidence and open-label treatment of interferon-induced major depressive disorder in patients with hepatitis C. Mol Psychiatry. 2002;7(9):942-7. doi: 10.1038/sj.mp.4001119. PMID 12399946
- [Background] Manns MP, McHutchison JG, Gordon SC, Rustgi VK, Shiffman M, Reindollar R, Goodman ZD, Koury K, Ling M, Albrecht JK. Peginterferon alfa-2b plus ribavirin compared with interferon alfa-2b plus ribavirin for initial treatment of chronic hepatitis C: a randomised trial. Lancet. 2001 Sep 22;358(9286):958-65. doi: 10.1016/s0140-6736(01)06102-5. PMID 11583749
- [Background] Pruessner JC, Wolf OT, Hellhammer DH, Buske-Kirschbaum A, von Auer K, Jobst S, Kaspers F, Kirschbaum C. Free cortisol levels after awakening: a reliable biological marker for the assessment of adrenocortical activity. Life Sci. 1997;61(26):2539-49. doi: 10.1016/s0024-3205(97)01008-4. PMID 9416776
- [Background] Speca M, Carlson LE, Goodey E, Angen M. A randomized, wait-list controlled clinical trial: the effect of a mindfulness meditation-based stress reduction program on mood and symptoms of stress in cancer outpatients. Psychosom Med. 2000 Sep-Oct;62(5):613-22. doi: 10.1097/00006842-200009000-00004. PMID 11020090
- [Background] Smyth JM, Stone AA, Hurewitz A, Kaell A. Effects of writing about stressful experiences on symptom reduction in patients with asthma or rheumatoid arthritis: a randomized trial. JAMA. 1999 Apr 14;281(14):1304-9. doi: 10.1001/jama.281.14.1304. PMID 10208146
- [Background] Teasdale JD, Scott J, Moore RG, Hayhurst H, Pope M, Paykel ES. How does cognitive therapy prevent relapse in residual depression? Evidence from a controlled trial. J Consult Clin Psychol. 2001 Jun;69(3):347-57. doi: 10.1037//0022-006x.69.3.347. PMID 11495165
- [Background] Valentine AD, Meyers CA, Kling MA, Richelson E, Hauser P. Mood and cognitive side effects of interferon-alpha therapy. Semin Oncol. 1998 Feb;25(1 Suppl 1):39-47. PMID 9482539
- [Background] Wichers M, Maes M. The psychoneuroimmuno-pathophysiology of cytokine-induced depression in humans. Int J Neuropsychopharmacol. 2002 Dec;5(4):375-88. doi: 10.1017/S1461145702003103. PMID 12466036